CLINICAL TRIAL: NCT06204341
Title: Towards Optimal Treatment for High Risk Prostate Cancer; Stereotactic Pelvic Radiotherapy with Focal Boost to the Primary Tumour
Brief Title: Towards Optimal Treatment for High Risk Prostate Cancer
Acronym: HYPOPRIME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haaglanden Medical Centre (Other)
Collaborators: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Leonard Bokhorst, MD, PhD, radiation oncologist, Haaglanden Medical Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P23.081
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-01

CONDITIONS: High Risk Prostate Carcinoma
Keywords: hypo fractionation; elective lymph node irradiation; focal boost; androgen deprivation therapy reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HYPOPRIME treatment (Experimental): Hypo fractionated pelvic radiotherapy with boost to primary tumour in the prostate with elective lymph node irradiation and minimized androgen deprivation therapy
  Interventions: Radiation: HYPOPRIME treatment

INTERVENTIONS:
Radiation: HYPOPRIME treatment — Hypo fractionated pelvic radiotherapy with boost to primary tumour in the prostate with elective lymph node irradiation and minimized androgen deprivation therapy

SUMMARY:
The goal of this clinical trial is to combine several optimized treatments of high risk prostate cancer. The main question to answer is: is it safe to combine these optimized treatments.

* patients will be irradiated on the prostate and (elective) lymph nodes more concentrated but with fewer hospital visits (hypofractionation)
* the tumor will get a higher dose
* androgen deprivation therapy will be reduced as much al possible preventing side effects

Researchers will compare oncological outcome and toxicity.

DETAILED DESCRIPTION:
Rationale: Recently several randomized trial have shown benefits of changes made to radiotherapy of (high risk) localized prostate cancer patients: A focal boost was shown to improve outcome in men with intermediate/high risk prostate cancer (FLAME trial). Elective lymph node irradiation was shown to improve outcome in high risk prostate cancer patients (POP-RT). (Extreme) hypo fractionation was shown to be safe for low/intermediate risk prostate cancer patients. In addition: the added benefit of ADT (with substantial toxicity) seems reduced with improvements made to treatment and diagnosis in recent years (DART 01/05); own recent work on this topic; to be published)). None off the above were combined into one ideal treatment for high risk prostate cancer.

Objective: Determine the safety (oncological outcome and toxicity) of an comprehensive treatment combining recent advances in the treatment of high risk prostate cancer.

Study design: prospective cohort study with matched contemporary control group Study population: Men with high risk prostate cancer with an indication for elective lymph node irradiation Intervention: hypo fractionated pelvic radiotherapy with boost to primary tumour in the prostate Main study parameters/endpoints: biochemical recurrence free survival and late toxicity Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The additional burden of the study is considered to be low, as additional tests or site visits in comparison to current clinical follow up are not planned. Regarding safety, different parts of the investigational treatment were already shown to be safe in previous studies. The current study aims to combine these different parts into one treatment. We estimate that the risks associated with combining these treatments are very limited.

ELIGIBILITY:
Inclusion Criteria:

* Men (aged ≥18 years of age) diagnosed within 6 months before inclusion with high risk prostate cancer:

  * T3 based on digital rectal examination AND/OR
  * Grade >= 4 AND/OR
  * PSA >=20 ug/L
* Indication for elective lymph node irradiation (based on current clinical guidelines) OR N1 on imaging (with a maximum of 4 suspect lymph nodes)

Exclusion Criteria:

* Prior pelvic radiotherapy
* TransUrethral Resection of the Prostate (TURP) < 3 months ago
* Prostatectomy or other primary treatment for prostate cancer (e.g. HIFU, cryotherapy, etc)
* contraindications to MRI
* no visible lesion on MRI in prostate for boost
* no PSMA-PET scan
* inflammatory bowel disease
* metastatic disease (M1)
* PSA >50
* unsuitable for SBRT or WPRT
* medical history of cancer other than basal cell carcinoma of the skin

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2032-12-18 (Estimated); Study Completion 2032-12-18 (Estimated)

PRIMARY OUTCOMES:
Biochemical recurrence free survival | 5 years
  rise of PSA 2 ng/ml above nadir
Late gastrointestinal and genito-urinary toxicity, and erectile dysfunction | at 6 months and 2 years
  according to CTC-AE v5

SECONDARY OUTCOMES:
Metastasis free survival | 5 years
  Metastasis free survival
Overall survival | 5 years
  Overall survival
Pattern of failure | 5 years
  based on PSMA in case of biochemical recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Leonard P Bokhorst, MD, PhD, Principal Investigator — Haaglanden Medical Centre
Locations (1):
- Haaglanden Medical Centre, Leidschendam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No